CLINICAL TRIAL: NCT01411384
Title: Evaluation of Corneal Hysteresis and Corneal Resistance Factor After Corneal Cross-linking for Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Georgios Labiris, Eye Institute of Thrace
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 20/21-07-2011
Record Dates: First submitted 2011-08-01; First posted 2011-08-08 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2011-07

CONDITIONS: Progressive Keratoconus
Keywords: Keratoconus (KC); Corneal collagen cross-linking (CXL); Corneal hysteresis (CH); Corneal resistance factor (CRF); Ocular Response Analyzer (ORA)
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Corneal collagen cross-linking — The same surgical procedure was applied to all keratoconus patients that included: Instillation of proparacaine hydrochloride 0.5% drops for topical anaesthesia, application of a sponge saturated with 10% alcohol to the central cornea for 30 seconds and subsequent de-epithelialization. Following de-epithelialization, a mixture of 0.1% riboflavin in 20% Dextran solution was instilled to the cornea for 30 minutes (2 drops every 2 minutes) prior to the irradiation, until the stroma was completely penetrated and aqueous was stained yellow. An 8.0mm diameter of central cornea was irradiated for 30 minutes by UVA light with a wavelength of 370nm and an irradiance of 3mW/cm2. Instillation of riboflavin drops (1 drop every 2 minutes) was continued during irradiation. Balanced salt solution (BSS) was applied every 6 minutes to moisten the cornea.
Device: Ocular Response Analyzer (ORA) — An air puff is released by a non-contact probe, which scanned the central area of the eye and send a signal to the ORA device. The air puff causes the cornea to move inward, past applanation, and into slight concavity. After milliseconds, the air pumps shut off, the pressure decreases, and the cornea begins to return in its normal state. The system monitors the entire process and measures two pressure values, which are determined from the inward and outward applanation processes. The aforementioned measuring procedure enables the determination of Corneal Hysteresis and Corneal Resistance Factor.

SUMMARY:
This study attempts to compare Corneal Hysteresis (CH) and Corneal Resistance Factor (CRF) in a series of keratoconic eyes before and after Corneal collagen cross-linking (CXL). Furthermore, among the objectives of the study is to reveal correlations between CH and CRF and a series of corneal indexes like the Corneal Thickness (CT), mean keratometry (Km) and corneal astigmatism (Astig).

The study adhered to the tenets of the Declaration of Helsinki and written informed consent was given by all participants. The study was conducted at the Eye Institute of Thrace (ΕΙΤ), in Alexandroupolis, Greece. EΙΤ is a Democritus University research institute focusing primarily on the conditions of the anterior segment of the eye.

Participants were recruited from the Outpatients Cornea service of the EIT in a consecutive if eligible basis. Fifty (50) eyes of thirty (30) patients with keratoconus were recruited for the sake of the study and formed the keratoconus group (KG). Eligible subjects for the keratoconus group had to present progressive keratoconus in consecutive corneal topographies, changes in refractive power, and deterioration of the visual acuity within a period of two years. Exclusion criteria included glaucoma, glaucoma suspicion, and intraocular pressure (IOP) lowering drugs administration. Further to glaucoma, exclusion criteria included central corneal thickness (CCT) less than 400μm, K-readings more than 60D, a history of herpetic keratitis, corneal scarring, severe eye dryness, pregnancy or nursing, current corneal infection, or underlying autoimmune disease.

Fifty (50) eyes of fifty (50) non-keratoconic, age-matched, individuals who visited our outpatient service formed the control group (CG). Further to keratoconus, and a spherical equivalent error above 3D, the same exclusion criteria applied to the control group members, as well. All participants wearing contact lenses were instructed to discontinue contact lens wear at least a month before measurements.

CRF and CH parameters were obtained while the patient was sitting on a chair in front of the Ocular Response Analyzer (ORA; Reichert Ophthalmic Instruments, Buffalo, NY, USA) device. Upon successful fixation of the patient's eye on a red blinking target, the operator activated the device. An air puff was released by a non-contact probe, which scanned the central area of the eye and sent a signal to the ORA. In brief, the air puff causes the cornea to move inward, past applanation, and into slight concavity. After milliseconds, the air pumps shut off, the pressure decreases, and the cornea begins to return in its normal state. The system monitors the entire process and measures two pressure values, which are determined from the inward and outward applanation processes. The aforementioned measuring procedure enables the determination of CH which is related to the viscoelastic structure of the corneal tissue, and is calculated as the difference between the two pressure values at the two applanation processes, and CRF which is indicative of the overall resistance of the cornea and is calculated as a linear function of the two pressures associated with the two applanation. In order to ensure accurate results, ORA was done four times for each eye, by the same operator. Signals that differ significantly in appearance from the other signals from the same eye were deleted.

The same surgical procedure was applied to all keratoconus patients that included: Instillation of proparacaine hydrochloride 0.5% drops for topical anaesthesia, application of a sponge saturated with 10% alcohol to the central cornea for 30 seconds and subsequent de-epithelialization by means of a hockey knife. Following de-epithelialization, a mixture of 0.1% riboflavin in 20% Dextran solution was instilled to the cornea for 30 minutes (2 drops every 2 minutes) prior to the irradiation, until the stroma was completely penetrated and aqueous was stained yellow. The ultraviolet A (UVA) radiation source that was used is UV-XTM (IROC AG, Zurich, Switzerland). In details, an 8.0mm diameter of central cornea was irradiated for 30 minutes by UVA light with a wavelength of 370nm and an irradiance of 3mW/cm2. Instillation of riboflavin drops (1 drop every 2 minutes) was continued during irradiation, as well, in order to sustain the necessary concentration of the riboflavin. Moreover, balanced salt solution (BSS) was applied every 6 minutes to moisten the cornea.

After treatment all patients were prescribed topical ofloxacin drops qid, fluorometholone qid and diclofenac nitrate qid, accompanied by frequent instillation of artificial tears. Soft therapeutic lens was applied until complete re-epithelialization of the cornea was detected. Follow up visits were performed on the 1st day, 7th day, 1st, 3rd, 6th and 12th month after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Progressive keratoconus in consecutive corneal topographies
* Changes in refractive power
* Deterioration of the visual acuity within a period of two years

Exclusion Criteria:

* Glaucoma
* Glaucoma suspicion
* Intraocular pressure lowering drugs administration
* Central Corneal Thickness less than 400μm
* K-readings more than 60D
* History of herpetic keratitis
* Corneal scarring
* Severe eye dryness
* Pregnancy
* Nursing
* Current corneal infection
* Underlying autoimmune disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Corneal Hysteresis (CH) | at 3rd, 6th and 12th month postoperatively
Change from baseline in Corneal Resistance Factor (CRF) | at 3rd, 6th and 12th month postoperatively

SECONDARY OUTCOMES:
Change from baseline in Average keratometry (Km) | at 3rd, 6th and 12th month postoperatively
Change from baseline in Corneal Thickness (CT) | at 3rd, 6th and 12th month postoperatively
Change from baseline in Corneal Astigmatism (Astig.) | at 3rd, 6th and 12th month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Democritus University